CLINICAL TRIAL: NCT04369807
Title: Mapping Organ Health Following COVID-19 Disease Due to SARS-CoV-2 Infection
Acronym: COVERSCAN
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: 20/SC/0185
Record Dates: First submitted 2020-04-22; First posted 2020-04-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: Metabolic Syndrome; Obesity; Fatty Liver Disease
MeSH Terms: conditions — COVID-19; Metabolic Syndrome; Obesity; Non-alcoholic Fatty Liver Disease | interventions — Genotype; Body Height; Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The tests consist of complete blood count (CBC), biochemical profile (e.g., electrolyte and renal panel, liver serum biochemistry) and stored serum/plasma.
  Genetic testing for genetic variants associated with this disease will also be carried out if the participant gives informed consent for genetic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Outpatient MRI — Participation in the study includes up to 3 visits to a partnering imaging facility - this will include measurement of height and weight (to calculate BMI), blood pressure measurement, 3 sets of blood tests, 3 Questionnaires and 3 MRI tests.
  There will be no medical interventions as part of the study. All participants will receive standard-of-care by their healthcare provider/s. With the participant's consent, the participant's primary care physician will be made aware of their participation in the study. Furthermore, participants will be informed of any structural abnormalities found in the MRI scan (e.g. abnormal vessels, haemangioma, tumour, cyst, among others) and abnormal blood test results as these may have clinical implications.
  Other Names: Outpatient blood tests for laboratory studies and genotyping; Outpatient measurements (height, weight, blood pressure); Online Questionnaires

SUMMARY:
A prospective, longitudinal, observational cohort study looking at patients following COVID-19 disease using multi-parametric magnetic resonance imaging (MRI) to assess the degree and prevalence of organ injury.

DETAILED DESCRIPTION:
To date, correctly, all of the Government's efforts have been dedicated to providing sufficient hospital space, and the appropriate equipment, for treating the most serious cases of COVID-19. Equally, enormous resource is being dedicated to developing technologies that determine who has the disease, and who has developed antibodies to it.

However, patients recovering from serious disease will also pose a huge, ongoing challenge. Not only are people with co-morbidities including underlying fatty liver disease, metabolic syndrome and diabetes at higher risk for complications with COVID-19; but patients discharged from hospital after severe COVID-19 are reported to have liver and kidney injuries, and impacts on pancreas and spleen. However, the extent of organ health/damage has not been mapped.

This is a prospective, longitudinal, observational cohort study looking at patients recovering from COVID-19 disease using multi-parametric magnetic resonance imaging (MRI) to assess the degree and prevalence of organ injury. This proposed study aims to measure the prevalence of organ volume changes and damage in lungs, heart, kidney, liver, pancreas, spleen as assessed by MRI among those having recovered, or recovering, from the SARS-CoV-2 infection - participants will have a final MRI scan at 12 months. Assessing the severity and sequelae of COVID-19 in patients is crucial to enable global planning for health-care needs. The study includes up to 3 visits for MRI scans and blood tests over a 12 month period. All participants will receive standard-of-care by their healthcare provider/s.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and older willing and able to give informed consent to participate in the study
* Recent confirmed diagnosis of SARS-CoV-2 RNA via a polymerase chain reaction (PCR) assay (having been discharged 7 or more days from hospital).

Exclusion Criteria:

* Symptoms of active respiratory viral infection:

  * high temperature (over 37.8C/100.04F)
  * cough (consistent for over an hour; 3 or more episodes in 24 hours)
* The participant may not enter the study with any known contraindication to magnetic resonance imaging (including but not limited to pregnancy, a pacemaker or other metallic unfixed implanted device, metallic fragments, extensive tattoos, severe claustrophobia).
* Any other cause, including a significant underlying disease or disorder which, in the opinion of the investigator, may put the participant at risk by participating in the study or limit the participant's ability to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recovered or recovering from COVID-19 disease, at least age 18 years and invited to partake in this study. Participants will previously have experienced symptomatic and confirmed COVID-19 disease and will be outpatients able to breath independently without oxygen. Participants will have been discharged back into the community with no respiratory symptoms for at least 7 days. Although subsequent negative testing for infectivity is ideal prior to study entry, participants will be considered non-infectious based on the absence of any fever or severe cough for at least 7 days, as per the advice of the UK Chief Medical Officer.
Sampling Method: Probability Sample
Enrollment: 693 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Characterise prevalence and severity of organ volume change and damage (heart, kidneys and liver) | 12 Months
  In patients recovering from COVID-19 disease:
  Characterise using summary statistics the prevalence and severity of organ volume change and damage to heart, kidneys and liver

SECONDARY OUTCOMES:
Characterise prevalence and severity of organ volume change and damage (lung, pancreas and spleen) | 12 Months
  In patients recovering from COVID-19 disease:
  To characterise using summary statistics the prevalence and severity of organ volume change and damage in lung, pancreas and spleen
Change from Baseline in liver-specific biomarkers: volume, iron corrected T1(cT1), fat content and T2star | 6 Months
  In patients recovering from COVID-19 disease:
  Characterise liver damage as assessed by liver volume in liters, iron corrected T1 (cT1) in milliseconds, liver fat content as %, liver T2star in milliseconds (a correlate of liver iron content)
Change from Baseline in organ-specific biomarkers characterising organ volume change in the heart and spleen along with organ volume and damage in the kidney, liver and pancreas assessed by volume, iron corrected T1 (cT1) and fat infiltration | 12 Months
  In patients recovering from COVID-19 disease:
  Characterise heart and spleen damage as assessed by liver volume in liters as well as kidney, liver and pancreas damage as assessed by volume in liters, iron corrected T1 (cT1) in milliseconds, fat infiltration as %, T2star in milliseconds (a correlate of liver iron content).
Change in patient reported outcome measured by the Dyspnea-12 questionnaire | 12 Months
  In patients recovering from COVID-19 disease:
  Change in patient reported outcome measures collected to assess breathlessness and its effect on overall health and daily life assessed by Dyspnea-12. Each question is assigned a value between: none, mild, moderate and severe and is used to assess breathing characteristics.
Change in patient reported outcome measured by the Saint George's Respiratory questionnaire (SGRQ) | 12 Months
  In patients recovering from COVID-19 disease:
  Change in patient reported outcome measures collected to assess breathlessness and its effect on overall health and daily life assessed by the St. George's Respiratory questionnaire. Each section comprises of questions in various formats allowing to assess which aspects of the illness cause the participant the most problems in daily life. There is no score on a scale to communicate the scale title.
Change in patient reported outcome measured by the EQ-5D-5L questionnaire | 12 Months
  In patients recovering from COVID-19 disease:
  Change in patient reported outcome measures collected to assess breathlessness and its effect on overall health and daily life assessed by the EQ-5D-5L questionnaire. Two main sections provide the opportunity to capture statements best describing a participant's daily health and a scale form 0 to 100 capturing self-reported health stats. (100 being the best health imaginable and vice versa)
Degree of change in liver MR-derived biomarkers | 12 Months
  In patients recovering from COVID-19 disease:
  Difference from Baseline in degree of change in liver MR-derived biomarkers with and without known genetic variants associated with liver disease (e.g., PNPLA3) using a paired t-test (or non-parametric alternative)

CONTACTS AND LOCATIONS:
Overall Officials: Rajarshi Banerjee, MSc, DPhil, Principal Investigator — Honorary Consultant Physician, Oxford University NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Mayo Clinic Healthcare, London
  - Gemini, Oxford

IPD SHARING:
Plan to Share IPD: No
Access to study data and/or results will be granted to Health Data Research UK (HDRUK), Public Health England (PHE) and to the World Health Organization (WHO).
  Furthermore, at the end of the study, the pooled and anonymous results of the questionnaires will be available to all participants upon their request. No individual participant will be identified.

REFERENCES:
- [Background] Bachtiar V, Kelly MD, Wilman HR, Jacobs J, Newbould R, Kelly CJ, Gyngell ML, Groves KE, McKay A, Herlihy AH, Fernandes CC, Halberstadt M, Maguire M, Jayaratne N, Linden S, Neubauer S, Banerjee R. Repeatability and reproducibility of multiparametric magnetic resonance imaging of the liver. PLoS One. 2019 Apr 10;14(4):e0214921. doi: 10.1371/journal.pone.0214921. eCollection 2019. PMID 30970039
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Bycroft C, Freeman C, Petkova D, Band G, Elliott LT, Sharp K, Motyer A, Vukcevic D, Delaneau O, O'Connell J, Cortes A, Welsh S, Young A, Effingham M, McVean G, Leslie S, Allen N, Donnelly P, Marchini J. The UK Biobank resource with deep phenotyping and genomic data. Nature. 2018 Oct;562(7726):203-209. doi: 10.1038/s41586-018-0579-z. Epub 2018 Oct 10. PMID 30305743
- [Background] Chen T, Wu D, Chen H, Yan W, Yang D, Chen G, Ma K, Xu D, Yu H, Wang H, Wang T, Guo W, Chen J, Ding C, Zhang X, Huang J, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical characteristics of 113 deceased patients with coronavirus disease 2019: retrospective study. BMJ. 2020 Mar 26;368:m1091. doi: 10.1136/bmj.m1091. PMID 32217556
- [Background] Cheng Y, Luo R, Wang K, Zhang M, Wang Z, Dong L, Li J, Yao Y, Ge S, Xu G. Kidney disease is associated with in-hospital death of patients with COVID-19. Kidney Int. 2020 May;97(5):829-838. doi: 10.1016/j.kint.2020.03.005. Epub 2020 Mar 20. PMID 32247631
- [Background] Ding Y, He L, Zhang Q, Huang Z, Che X, Hou J, Wang H, Shen H, Qiu L, Li Z, Geng J, Cai J, Han H, Li X, Kang W, Weng D, Liang P, Jiang S. Organ distribution of severe acute respiratory syndrome (SARS) associated coronavirus (SARS-CoV) in SARS patients: implications for pathogenesis and virus transmission pathways. J Pathol. 2004 Jun;203(2):622-30. doi: 10.1002/path.1560. PMID 15141376
- [Background] Driggin E, Madhavan MV, Bikdeli B, Chuich T, Laracy J, Biondi-Zoccai G, Brown TS, Der Nigoghossian C, Zidar DA, Haythe J, Brodie D, Beckman JA, Kirtane AJ, Stone GW, Krumholz HM, Parikh SA. Cardiovascular Considerations for Patients, Health Care Workers, and Health Systems During the COVID-19 Pandemic. J Am Coll Cardiol. 2020 May 12;75(18):2352-2371. doi: 10.1016/j.jacc.2020.03.031. Epub 2020 Mar 19. PMID 32201335
- [Background] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Gurwitz D. Angiotensin receptor blockers as tentative SARS-CoV-2 therapeutics. Drug Dev Res. 2020 Aug;81(5):537-540. doi: 10.1002/ddr.21656. Epub 2020 Mar 4. PMID 32129518
- [Background] Harrison SA, Bashir MR, Guy CD, Zhou R, Moylan CA, Frias JP, Alkhouri N, Bansal MB, Baum S, Neuschwander-Tetri BA, Taub R, Moussa SE. Resmetirom (MGL-3196) for the treatment of non-alcoholic steatohepatitis: a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2019 Nov 30;394(10213):2012-2024. doi: 10.1016/S0140-6736(19)32517-6. Epub 2019 Nov 11. PMID 31727409
- [Background] Harrison SA, Rossi SJ, Paredes AH, Trotter JF, Bashir MR, Guy CD, Banerjee R, Jaros MJ, Owers S, Baxter BA, Ling L, DePaoli AM. NGM282 Improves Liver Fibrosis and Histology in 12 Weeks in Patients With Nonalcoholic Steatohepatitis. Hepatology. 2020 Apr;71(4):1198-1212. doi: 10.1002/hep.30590. Epub 2019 Apr 10. PMID 30805949
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Pavlides M, Banerjee R, Sellwood J, Kelly CJ, Robson MD, Booth JC, Collier J, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging predicts clinical outcomes in patients with chronic liver disease. J Hepatol. 2016 Feb;64(2):308-315. doi: 10.1016/j.jhep.2015.10.009. Epub 2015 Nov 10. PMID 26471505
- [Background] Pavlides M, Banerjee R, Tunnicliffe EM, Kelly C, Collier J, Wang LM, Fleming KA, Cobbold JF, Robson MD, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging for the assessment of non-alcoholic fatty liver disease severity. Liver Int. 2017 Jul;37(7):1065-1073. doi: 10.1111/liv.13284. Epub 2017 May 30. PMID 27778429
- [Background] Verity R, Okell LC, Dorigatti I, Winskill P, Whittaker C, Imai N, Cuomo-Dannenburg G, Thompson H, Walker PGT, Fu H, Dighe A, Griffin JT, Baguelin M, Bhatia S, Boonyasiri A, Cori A, Cucunuba Z, FitzJohn R, Gaythorpe K, Green W, Hamlet A, Hinsley W, Laydon D, Nedjati-Gilani G, Riley S, van Elsland S, Volz E, Wang H, Wang Y, Xi X, Donnelly CA, Ghani AC, Ferguson NM. Estimates of the severity of coronavirus disease 2019: a model-based analysis. Lancet Infect Dis. 2020 Jun;20(6):669-677. doi: 10.1016/S1473-3099(20)30243-7. Epub 2020 Mar 30. PMID 32240634
- [Background] Wang T, Du Z, Zhu F, Cao Z, An Y, Gao Y, Jiang B. Comorbidities and multi-organ injuries in the treatment of COVID-19. Lancet. 2020 Mar 21;395(10228):e52. doi: 10.1016/S0140-6736(20)30558-4. Epub 2020 Mar 11. No abstract available. PMID 32171074
- [Background] Xu L, Liu J, Lu M, Yang D, Zheng X. Liver injury during highly pathogenic human coronavirus infections. Liver Int. 2020 May;40(5):998-1004. doi: 10.1111/liv.14435. Epub 2020 Mar 30. PMID 32170806
- [Background] Zhang C, Shi L, Wang FS. Liver injury in COVID-19: management and challenges. Lancet Gastroenterol Hepatol. 2020 May;5(5):428-430. doi: 10.1016/S2468-1253(20)30057-1. Epub 2020 Mar 4. No abstract available. PMID 32145190
- [Result] Dennis A, Cuthbertson DJ, Wootton D, Crooks M, Gabbay M, Eichert N, Mouchti S, Pansini M, Roca-Fernandez A, Thomaides-Brears H, Kelly M, Robson M, Hishmeh L, Attree E, Heightman M, Banerjee R, Banerjee A. Multi-organ impairment and long COVID: a 1-year prospective, longitudinal cohort study. J R Soc Med. 2023 Mar;116(3):97-112. doi: 10.1177/01410768231154703. Epub 2023 Feb 14. PMID 36787802
- [Result] Roca-Fernandez A, Dennis A, Nicholls R, McGonigle J, Kelly M, Banerjee R, Banerjee A, Sanyal AJ. Hepatic Steatosis, Rather Than Underlying Obesity, Increases the Risk of Infection and Hospitalization for COVID-19. Front Med (Lausanne). 2021 Mar 29;8:636637. doi: 10.3389/fmed.2021.636637. eCollection 2021. PMID 33855033
- [Result] Davis HE, McCorkell L, Vogel JM, Topol EJ. Long COVID: major findings, mechanisms and recommendations. Nat Rev Microbiol. 2023 Mar;21(3):133-146. doi: 10.1038/s41579-022-00846-2. Epub 2023 Jan 13. PMID 36639608
- [Result] Roca-Fernandez A, Wamil M, Telford A, Carapella V, Borlotti A, Monteiro D, Thomaides-Brears H, Kelly M, Dennis A, Banerjee R, Robson M, Brady M, Lip GYH, Bull S, Heightman M, Ntusi N, Banerjee A. Cardiac abnormalities in Long COVID 1-year post-SARS-CoV-2 infection. Open Heart. 2023 Feb;10(1):e002241. doi: 10.1136/openhrt-2022-002241. PMID 36822818
- [Result] Borlotti A, Thomaides-Brears H, Georgiopoulos G, Banerjee R, Robson MD, Fusco DN, Masci PG. The Additive Value of Cardiovascular Magnetic Resonance in Convalescent COVID-19 Patients. Front Cardiovasc Med. 2022 Apr 7;9:854750. doi: 10.3389/fcvm.2022.854750. eCollection 2022. PMID 35463767
- [Result] Dennis A, Wamil M, Alberts J, Oben J, Cuthbertson DJ, Wootton D, Crooks M, Gabbay M, Brady M, Hishmeh L, Attree E, Heightman M, Banerjee R, Banerjee A; COVERSCAN study investigators. Multiorgan impairment in low-risk individuals with post-COVID-19 syndrome: a prospective, community-based study. BMJ Open. 2021 Mar 30;11(3):e048391. doi: 10.1136/bmjopen-2020-048391. PMID 33785495
- See also: WHO. (2020, February 28). Report of the WHO-China Joint Mission on Coronavirus Disease (COVID-19). — https://www.who.int/docs/default-source/coronaviruse/who-china-joint-mission-on-covid-19-final-report.pdf
- See also: Parisinos CA, W. H. (2020). Genetic studies of magnetic resonance imaging of the liver implicate metal ion transporters in the pathogenesis of steatohepatitis in UK Biobank. J Hepatol — https://pubmed.ncbi.nlm.nih.gov/32247823/
- See also: COVID-19 Surveillance Group. (2020). Characteristics of COVID-19 patients dying in Italy: report based on available data on March 20th, 2020. : ; 2020. Rome, Italy: Instituto Superiore Di Sanita. — https://www.epicentro.iss.it/coronavirus/bollettino/Report-COVID-2019
- See also: Mapping Organ Health following COVID-19 Disease due to SARS-CoV-2 infection — https://www.perspectum.com/for-researchers